CLINICAL TRIAL: NCT06460090
Title: Evaluating a Targeted Selective Speech, Language, and Communication Intervention at Scale - Protocol for the 'Happy Talk' Cluster Randomised Controlled Trial.
Acronym: HappyTalk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DIFA-2023-001; DIFA-2023-001 (Other Grant/Funding Number: Health Research Board, Ireland)
Record Dates: First submitted 2024-05-20; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Developmental Language Disorder and Language Impairment; Deprivation
Keywords: Developmental language disorder; social disadvantage; public health; intervention; children; speech and language
MeSH Terms: conditions — Language Development Disorders; Language Disorders; Speech; Language

STUDY DESIGN:
Intervention Model Description: The design is a parallel cluster randomised trial of a 12-week manualised intervention delivered in pre/school settings serving socially disadvantaged communities, over two academic years in Ireland. Following baseline data and scoring, randomization will take place at the level of the setting whereby pre/schools will be allocated to either a treatment or a "business as usual" control group, stratified for geographical region.
Who Masked: Investigator, Outcomes Assessor
Masking Description: All outcomes will be administered blind and the investigator team analysing parent videos will be blind to time and treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): The intervention has two components, parent and preschool. The parent component includes twelve 1-hour sessions delivered in two 30-min units, over the three terms of the preschool year (in 4 week blocks). For the first 30 min, parents engage in group training with the SLT in a room within the preschool, in which they are introduced to language promoting strategies and techniques. This is followed by 30 min of coaching, with parents practising their newly acquired skills, with their children in the preschool.
  The preschool component is made up of 4 workshops. The first takes place in each preschool before the 12-week parent programme begins and the remaining three take place following each 4-week parent intervention block. Workshops focus on core interaction skills covered with parents as well as literacy skills and phonological awareness skills. Staff also get the opportunity to practice their skills and engage in coaching.
  Interventions: Behavioral: Happy Talk
- Usual Care (No Intervention): Usual care is the Early Childhood care and Education programme (ECCE) for preschool. The programme is provided for three hours per day, five days per week over 38 weeks per year. Childcare services taking part in the programme provide a pre-school educational programme which adheres to the principles of Síolta, the national framework for early years care and education. The most commonly implemented programme is 'Aistear' which is based on 12 principles of early learning and development, presented in three groups 1) children and their lives in early childhood 2) children's connections with others and 3) how children learn and develop. Communication and language is one element of the third component.
  Junior infants is the first year of an 8 year cycle in primary education. The primary curriculum is presented in 7 areas: Art; Mathematics, Social Environmental and Scientific Education; Physical Education; Religious Education; Primary Language; and Social, personal and Health Education.

INTERVENTIONS:
Behavioral: Happy Talk — A targeted selective speech language and communication programme embedded in the community, designed for people livling in social disadvantage.
  Arms: Intervention arm

SUMMARY:
The overall aim of this clinical trial is to evaluate an at scale version of 'Happy Talk' in a large scale effectiveness study (examining inputs, outputs and outcomes) based on a sample of children from socially disadvantaged areas. Researchers will compare Happy Talk to usual care and children's allocation to the programme will be decided on randomly.

The investigators also aim to

* complete a pre-trial process evaluation to inform intervention implementation - examining factors which promote parental engagement and partnership between SLTs and educators and incorporating these into SLT training and future rollouts of the programme.
* complete a concurrent process evaluation from a realist perspective to examine how the mechanisms underpinning Happy Talk are influenced by the implementation context and therefore what would need to be considered for successful implementation across varied settings. Our SWAT is embedded in this process evaluation and addresses the Trials Methodology Research Network methodological priority questions 1 and 5 https://priorityresearch.ie/priority-one-questions/
* Complete an economic evaluation in which compare the costs and benefits of Happy Talk are compared to standard pre/school care.

The study aims to answer the following research questions:

When implemented at scale

1. Does 'Happy Talk', a targeted selective intervention focused on increasing parent and early educator responsive interaction, improve language and quality of-life (QoL) outcomes in socially disadvantaged preschool and young school-aged children?
2. Does Happy Talk enhance responsiveness and language promoting behaviours in home and pre/school contexts?
3. What programme features support successful real-world application of 'Happy Talk' including factors which promote parental engagement; partnership between SLTs and educators; and fidelity of implementation?
4. How do contextual factors influence Happy Talk implementation /outcomes?
5. How can trials become part of routine care?
6. Is Happy Talk cost effective compared to usual care?

Intervention: The programme is informed by general systems theory and is embedded in the preschools, and homes of socially disadvantaged children with the aim of effecting change in parent and educator behaviour. There are both parent and preschool staff components to the programme.

ELIGIBILITY:
Inclusion Criteria for pre/schools:

* Those falling within the Health Services Executive Community Healthcare Organisation (CHO) area for which support has been offered.
* Those attached to DEIS schools (Delivering Equality of Opportunity in Schools i.e., those including a high concentration of students from socioeconomically disadvantaged backgrounds)
* Child and Family Resource centres (established in Ireland for children from disadvantaged backgrounds)

Exclusion Criteria:

* Pre/schools outside of supported areas.
* Schools that are not defined as DEIS schools.
* Preschools not attached to DEIS schools.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 840 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Expressive and receptive language on the standardised Preschool Language Scale 5 (PLS-5) | The measure will be completed at baseline, immediately post the 12 week intervention and 6 months post-intervention.
  This is a standardized norm referenced language assessment that yields standard scores for total language, auditory comprehension, and expressive communication. A standard score of 100 represents the performance of a typical child at a given age, the higher the standard score the better the performance. Standard scores between 85 and 115 correspond to one standard deviation below and above the mean, respectively; scores within this range are considered to be within normal limits.
Focus on the Outcomes of Communication Under Six (FOCUS) | The measure will be completed at baseline, immediately post the 12 week intervention and 6 months post-intervention.
  The Focus on the outcomes of communication under 6 (FOCUS-34) is a clinical tool designed to evaluate change in communicative-participation in preschool children. The parent form consists of 34 statements - aimed at taking a snapshot of children's skills as they are on that day. Parents are asked to rate each statement using a 7 point scale, ranging from 'not at all like my child' to 'exactly like my child'. This yields a total score ranging from 50 to 350 with a higher score indicating a better outcome.

SECONDARY OUTCOMES:
Parent - Maternal Responsive Behaviours Coding Scheme (MRBCS) | The measure will be completed at baseline, immediately post the 12 week intervention and 6 months post-intervention.
  The Maternal Responsive Behaviours Coding Scheme (MRBCS - Levickis et al. 2014) is an observational coding scheme of parent- child interaction. Implementation of the MRBCS yields a total number of occurrences of one of four parental responsive behaviours (Expansions; Imitations; Responsive Questions; and Labels), for a given period. By summing the frequency scores for each behaviour, an overall score of parental responsiveness can be calculated. The lowest score is 0 and the highest score is not specified. The higher the score the greater the number of parental responsive behaviours - yielding better outcomes.
Child - Paediatric Quality of Life Inventory (PedsQL) Parent report for Toddlers | Quality of life measures will be completed at baseline, immediately post the 12 week intervention and 6 months post-intervention.
  This is a parent proxy-report scale of health-related QoL in young children. The PedsQL for toddlers contains 21 items and measures four health dimensions: physical, emotional, social, and school functioning (questions related to school or daycare if attended). The tool asks, "please tell us how much of a problem each item has been for your child during the past one month." Parents are required to rate each item on a scale of 0- 4 (0 indicating never a problem and 4 almost always a problem). The ratings are tallied yielding a total score for each section, the higher score indicating a greater level of difficulty.
Setting - Classroom assessment scoring system (CLASS). | The measure will be completed at baseline, immediately post the 12 week intervention and 6 months post-intervention.
  The Classroom Assessment Scoring System (Pianta, La Paro, & Hamre, 2008) is a theoretically-based and empirically-supported observation instrument designed to assess the quality of interactions between teachers and students in the classroom. The CLASS measures three broad domains of teacher-student interactions: Emotional Support, Classroom Organization, and Instructional Support. These three domains are comprised of 10 specific dimensions of teacher-student interactions. Assessors assign scores to classrooms on each of the 10 dimensions on a 7-point scale.
Child - Child Health Utility Instrument (CHU9D). | The measure will be completed at baseline, immediately post the 12 week intervention and 6 months post-intervention.
  This is a parent proxy-report scale of health related quality of life in young children. The CHU9D for children < 5years) consists of 11 questions and parents are asked to base their responses on how their child is feeling on the day of completion. It consists of a descriptive system and a set of preference weights, which give utility values for each health state described by the descriptive system, allowing the calculation of QALYs.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Frizelle, Principal Investigator — University College Cork
Locations (4):
- Ireland (4):
  - Dublin North West, Dublin
  - Galway, Galway
  - Wexford, Wexford
  - Wicklow, Wicklow

IPD SHARING:
Plan to Share IPD: Yes
Electronic Data Capture platform (Castor EDC) will be used throughout this project.
  Data sharing and preservation: Data sharing repositories will be formerly identified via careful alignment of the expected data object outputs and evaluated using the re3data resource. This is to ensure maximum utility and interoperability of the final data package(s) and assignment of a persistent digital object identifier (DOI). Additional post-study data provenance will be enacted through sharing of analysis scripts and study protocols via Open Science Framework and/or the HRB Open Research platform projects with accompanying DOI(s). Study findings will be written up as journal publications, and published open access.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available when the study is completed.
Access Criteria: All study information will be submitted to an open science repository.

REFERENCES:
- [Background] Frizelle P, Mullane E, O'Shea A, Ceroni A, Dahly D, Horgan A, Levickis P, Mckean C. Happy Talk: A pilot effectiveness study of a targeted-selective speech-language and communication intervention for children from areas of social disadvantage. Int J Lang Commun Disord. 2021 Sep;56(5):954-974. doi: 10.1111/1460-6984.12648. Epub 2021 Jul 28. PMID 34322955
- [Background] Frizelle P, Mckean C, O'Shea A, Horgan A, Murphy A. Economic evaluation of the Happy Talk pilot effectiveness trial: A targeted selective speech, language and communication intervention for children from areas of social disadvantage. Int J Speech Lang Pathol. 2022 Apr;24(2):200-211. doi: 10.1080/17549507.2021.1975815. Epub 2021 Sep 20. PMID 34543137
- [Derived] Frizelle P, O'Shea A, Murphy A, Dahly D, McKean C. Evaluating a targeted selective speech, language, and communication intervention at scale - Protocol for the Happy Talk cluster randomised controlled trial. HRB Open Res. 2025 Jan 31;7:65. doi: 10.12688/hrbopenres.13973.3. eCollection 2024. PMID 39931387